CLINICAL TRIAL: NCT00315419
Title: Screening Protocol and Longitudinal Study of Bone Marrow Failure Syndromes and Cytopenias
Brief Title: Identifying Characteristics of Bone Marrow Failure Syndromes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Office of Rare Diseases (ORD) (NIH)
Collaborators: Rare Diseases Clinical Research Network (Network)
Responsible Party: Jaroslaw Maciejewski, MD, PhD, Cleveland Clinic Foundation
Other Study IDs: RDCRN 5401; RR19397-03
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2009-07

CONDITIONS: Bone Marrow Failure Syndromes; Anemia, Aplastic; Myelodysplastic Syndromes; Hemoglobinuria, Paroxysmal; Red-Cell Aplasia, Pure; Purpura, Thrombocytopenic; Leukemia, Lymphocytic
Keywords: Large Granular Lymphocyte Leukemia; Amegakaryocytic Thrombocytopenic Purpura; Idiopathic Pure Red Cell Aplasia; Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Bone Marrow Failure Disorders; Anemia, Aplastic; Myelodysplastic Syndromes; Hemoglobinuria, Paroxysmal; Red-Cell Aplasia, Pure; Purpura, Thrombocytopenic; Leukemia, Lymphoid; Leukemia, Large Granular Lymphocytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual samples from peripheral blood and bone marrow aspiration/biopsies

SUMMARY:
Bone marrow failure syndromes (BMFS) are rare disorders characterized by dysfunctional hematopoietic stem cells, which give rise to all red and white blood cells. The deficiency of blood cells, or cytopenia, caused by this malfunction leads to an assortment of diseases and disorders, all of which are characterized as BMFS. Because these diseases are rare, conducting research on them is difficult, and standards of treatment for most BMFS have yet to be developed. This study will collect clinical and laboratory data from people with BMFS to identify the characteristics and biological markers associated with these diseases over time. This information will assist doctors and researchers to develop better therapies and diagnostic tests that will help improve the management of BMFS and cytopenias.

DETAILED DESCRIPTION:
BMFS result from hematopoietic progenitor or stem cell failure within the bone marrow. Specific causes of this problem, however, have been difficult to identify, as BMFS occur sporadically. For the same reason, few studies have been conducted to find out more about these diseases and to develop more appropriate and effective therapies. Aplastic anemia (AA) is the most common of all BMFS. Other types of BMFS include the following: myelodysplastic syndrome (MDS); paroxysmal nocturnal hemoglobinuria (PNH); pure red cell aplasia (PRCA); amegakaryocytic thrombocytopenic purpura (ATP); and large granular lymphocyte leukemia (LGL leukemia). Though AA is the most common of the BMFS, all BMFS are closely related in terms of their symptoms and characteristics. This study will collect clinical and laboratory data from people with BMFS to identify the characteristics and biological markers specific to each disease as it evolves. This information will assist doctors and researchers to devise better therapies and diagnostic tests that will help improve the management of BMFS and cytopenias.

Participants in this observational study will report to the study site for an initial screening visit, followed by study visits every 6 months for at least 5 years. At each visit, participants will be interviewed and examined by a physician. Laboratory tests, including blood collection and a bone marrow aspirate, will also be performed. Data collected for this study's database will be used to determine the prevalence of clinical events and laboratory abnormalities over the course of disease, to study the evolution of disease parameters and symptoms, and to evaluate current therapies and diagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the following diseases: aplastic anemia; myelodysplastic syndrome; paroxysmal nocturnal hemoglobinuria; idiopathic pure red cell aplasia; amegakaryocytic thrombocytopenia purpura; or large granular lymphocyte leukemia

Exclusion Criteria:

* N/A

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with bone marrow failure syndromes
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw P. Maciejewski, MD, PhD, Study Chair — The Cleveland Clinic
Locations (4):
- United States (4):
  - University of California, Los Angeles, Department of Hematology and Oncology, Los Angeles, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Pennsylvania State University Cancer Center, Hershey, Pennsylvania

REFERENCES:
- [Background] Young NS. Immunosuppressive treatment of acquired aplastic anemia and immune-mediated bone marrow failure syndromes. Int J Hematol. 2002 Feb;75(2):129-40. doi: 10.1007/BF02982017. PMID 11939258
- [Background] Plasilova M, Risitano A, Maciejewski JP. Application of the molecular analysis of the T-cell receptor repertoire in the study of immune-mediated hematologic diseases. Hematology. 2003 Jun;8(3):173-81. doi: 10.1080/1024533031000107505. PMID 12745651
- [Background] Frickhofen N, Heimpel H, Kaltwasser JP, Schrezenmeier H; German Aplastic Anemia Study Group. Antithymocyte globulin with or without cyclosporin A: 11-year follow-up of a randomized trial comparing treatments of aplastic anemia. Blood. 2003 Feb 15;101(4):1236-42. doi: 10.1182/blood-2002-04-1134. Epub 2002 Oct 10. PMID 12393680
- [Background] Molldrem JJ, Leifer E, Bahceci E, Saunthararajah Y, Rivera M, Dunbar C, Liu J, Nakamura R, Young NS, Barrett AJ. Antithymocyte globulin for treatment of the bone marrow failure associated with myelodysplastic syndromes. Ann Intern Med. 2002 Aug 6;137(3):156-63. doi: 10.7326/0003-4819-137-3-200208060-00007. PMID 12160363
- [Background] Sloand E, Kim S, Maciejewski JP, Tisdale J, Follmann D, Young NS. Intracellular interferon-gamma in circulating and marrow T cells detected by flow cytometry and the response to immunosuppressive therapy in patients with aplastic anemia. Blood. 2002 Aug 15;100(4):1185-91. doi: 10.1182/blood-2002-01-0035. PMID 12149196